CLINICAL TRIAL: NCT04513496
Title: Delivery of HIV Care Through Telemedicine in Public Hospitals in Buenos Aires, Argentina During COVID-19 Pandemic: Implementation Research
Brief Title: Telemedicine in HIV Care in Buenos Aires
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundacion Ibis (Other)
Responsible Party: Sponsor
Other Study IDs: TM HIV BA
Record Dates: First submitted 2020-08-04; First posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Telemedicine; HIV-1-infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this investigation is to conduct an implementation research to facilitate and evaluate the implementation of VCT((Videoconsult through telemedicine) among HIV HCP(healthcare providers) and PLWH(people living with HIV)

DETAILED DESCRIPTION:
Through prospective observational methodology the investigators are planning to evaluate VCT(Videoconsult through telemedicine) implementation. Both quantitative and qualitative analysis (mixed methods) will take part in the assessment. Quantitative data will be useful to obtain objective data in terms of proportion of subjects using the intervention, adoption by health care workers and measuring effectiveness. Additionally, qualitative methods will help to understand the outcomes focusing on the barriers and facilitators from both the HCW and patients, and their feedback on continuous implementation.

Hence, perceptions of a vast group of patients and HCW will take a critical point in the qualitative analysis. Finally, by evidencing effectiveness, the investigators will be able to generalize and maintain this intervention as a good clinical practice. Due to the scope of the outcomes, the investigators will use RE-AIM framework.

ELIGIBILITY:
Inclusion Criteria:

* 18 years-old or older
* Access to internet
* Willing to participate

Exclusion Criteria:

* do not understand the purpose and study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PLWH(people living with HIV) that receive care in Buenos Aires public hospitals
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Telemedicine Reach. RE-AIM framework | 18 months
  Proportion of included patients over all patients eligible
Telemedicine Effectiveness. RE-AIM framework | 18 months
  Proportion of treatment interruptions and undetectable HIV viral load
Telemedicine Adoption. RE-AIM framework | 18 months
  Proportion of physicians adopting VC, barriers and facilitators to adopt telemedicine
Telemedicine Implementation.RE-AIM framework | 18 months
  Time and cost needed to deliver the intervention
Telemedicine Manteinance. RE-AIM framework | 18 months
  Inclusion of VCT into routine activity, Satisfaction of HCP(healthcare proffesionals and patients with videoconsultation